CLINICAL TRIAL: NCT04942886
Title: A Randomized, Prospective, Comparative Study of the Effectiveness of Prophylactic Entecavir Treatment for HBV Reactivation in Past HBV Infected Patients With Hematopoietic Stem Cell Transplantation
Brief Title: Prophylactic Entecavir for HBV Reactivation in Past HBV Infected Patients With Hematopoietic Stem Cell Transplantation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Dong-Gun Lee, professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC20MISI0622
Record Dates: First submitted 2021-06-15; First posted 2021-06-29 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hepatitis B Reactivation; Hematopoietic Stem Cell Transplantation; Antiviral Drug; HBV
Keywords: Hepatitis B Reactivation; hematopoietic stem cell transplantation; Prophylatic antiviral agents; Past HBV infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The intervention group take entecavir 0.5mg everyday by oral administration for 3 years after allogeneic hematopoietic stem cell transplantation. The intervention group visit clinic every month and examined liver function test, HBsAg/Ab. HBV DNA level is examined at every 3 months.
  Interventions: Drug: Baracle Tab.®
- delayed treatment group (No Intervention): The delayed treatment group (control group) visit clinic every month and examined liver function test, HBsAg/Ab for 3 years after allogeneic hematopoietic stem cell transplantation. HBV DNA level is examined at every 3 months for 3 years after allogenic hematopoietic stem cell transplantation. If the patient in the delayed treatment group shows HBV reactivation (positive HBsAg or HBV DNA ≥10 IU/mL), entecavir treatment is started.

INTERVENTIONS:
Drug: Baracle Tab.® — The intervention group take entecavir 0.5mg everyday by oral administration for 3 years after hematopoietic stem cell transplantation.
  Other Names: Prophylactic treatment group
  Arms: Treatment group

SUMMARY:
This study is a randomized, prospective, comparative study of the effectiveness of prophylactic entecavir treatment for HBV reactivation in past HBV infected patients (HBsAg-, HBcIgG+) with allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
This study is a randomized, prospective, comparative study of the effectiveness of prophylactic entecavir treatment for HBV reactivation in past HBV infected patients (HBsAg-, HBcIgG+) with allogeneic hematopoietic stem cell transplantation.

In this study, patients are randomized into treatment group or delayed treatment group.

* Stratified randomization (Block randomization within strata) according to the presence of HBsAb at baseline was used in this study.

1. Experimental: Treatment group (n=113) The intervention group take entecavir 0.5mg everyday by oral administration for 3 years after allogeneic hematopoietic stem cell transplantation. The intervention group visit clinic every month and examined liver function test, HBsAg/Ab. HBV DNA level is examined at every 3 months.

   * oral administration of entecavir is planned to start within 7 days after hematopoietic stem cell transplantation.
2. No Intervention: delayed treatment group (n=113) The delayed treatment group visit clinic every month and examined liver function test, HBsAg/Ab. HBV DNA level is examined at every 3 months. If the patient in the delayed treatment group shows HBV reactivation (positive HBsAg or HBV DNA ≥10 IU/mL), entecavir treatment is started.

ELIGIBILITY:
1. Inclusion Criteria:

   * Age: 19 - 70
   * Patients receiving allogeneic hematopoietic stem cell transplantation
   * HBV serologic test: HBsAg (-), anti-HBc IgG (+) before receiving allogeneic hematopoietic stem cell transplantation
   * ECOG performence: 0-2
   * patients with informed consent
2. Exclusion Criteria:

   * HBV DNA (+, ≥10 IU/mL) at the time of screening
   * Receiving hematopoietic stem cell transplantation from donor with HBsAg+
   * Combined other chronic liver disease (severe alcoholics, autoimmune hepatitis, chronic hepatitis C etc.)
   * HIV (+)
   * Previous antiviral therapy history for chronic hepatitis B
   * Other concomitant malignancy
   * Combined autoimmune disease (rheumatic arthritis, SLE etc)
   * CTP class B, C
   * Decompensated complications (ascites, hepatic encephalopathy etc.)
   * Active tuberculosis
   * Patients with lymphoma
   * Patients receiving autologous hematopoietic stem cell transplantation

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the rate of HBV reactivation between the treatment and delayed treatment groups. | The primary outcome is evaluated during 3 years after hematopoietic stem cell transplantation
  Comparing the rate of HBV reactivation between the treatment and delayed treatment groups during 3 years after hematopoietic stem cell transplantation
  * Definition of HBV reactivation: HBsAg ≥ 1.0 S/CO or HBV DNA ≥ 10 IU/mL

SECONDARY OUTCOMES:
Comparison of the rate of active hepatitis with HBV reactivation between the treatment and delayed treatment groups. | The secondary outcomes are evaluated during 3 years after hematopoietic stem cell transplantation.
  Comparing the rate of active hepatitis with HBV reactivation between the treatment and delayed treatment groups.
  * Definition of active hepatitis: ALT >= 2 times of upper normal limit
Comparison of the rate of hepatic failure related to HBV reactivation between the treatment and delayed treatment groups. | The secondary outcomes are evaluated during 3 years after hematopoietic stem cell transplantation.
  Comparing the rate of hepatic failure between the treatment and delayed treatment groups.
Comparison of the rate of survival related to HBV reactivation between the treatment and delayed treatment groups. | The secondary outcomes are evaluated during 3 years after hematopoietic stem cell transplantation.
  Comparing the rate of survival related to HBV reactivation between the treatment and delayed treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Won Jang, Professor, Study Chair — Seoul St. Mary's Hospital, the catholic university of Korea
Locations (1):
- Jeong Won Jang, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
According to the guideline of our institutional review board, the patient data could not be opened to other researchers.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT04942886/Prot_SAP_001.pdf